CLINICAL TRIAL: NCT03319823
Title: A Pilot Study: Treating Nocturnal Hypertension and Nocturia in African American Men
Brief Title: Treating Nocturnal Hypertension and Nocturia in African American Men
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the Pandemic, we decided to end this study.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Florian Rader, Co-Director, Clinic for Hypertrophic Cardiomyopathy and Aortopathies, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 48809
Record Dates: First submitted 2017-10-10; First posted 2017-10-24 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Study Design and Procedures
  Participants who meet the inclusion criteria will be contacted by the study team. The purpose of the study will be explained, and they will be asked to sign an informed consent form. Based on their nocturnal systolic blood pressure, the investigators will assign participants to one of two treatment groups:
  * Group (1): Thiazide Therapy Group: Men without diabetes, and mild hypertension - a sleeping systolic blood pressure of 125-139 mm Hg, and an awake average blood pressure of < 160 mm Hg.
  * Group (2): Combination Therapy Group: Men with diabetes, or with more severe hypertension - a sleeping blood pressure of ≥ 140 mm Hg, or an awake average blood pressure of ≥ 160 mm Hg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Thiazide Therapy Group (Experimental): • Group (1): Thiazide Therapy Group: Men without diabetes, and mild hypertension - a sleeping systolic blood pressure of 125-139 mm Hg, and an awake average blood pressure of < 160 mm Hg
  Interventions: Drug: Thiazide Treatment Group; Drug: Intensified Thiazide Treatment Group
- Combination Therapy Group (Experimental): • Group (2): Combination Therapy Group: Men with diabetes, or with more severe hypertension - a sleeping blood pressure of ≥ 140 mm Hg, or an awake average blood pressure of ≥ 160 mm Hg.
  Interventions: Drug: Combination Medication Treatment Group

INTERVENTIONS:
Drug: Thiazide Treatment Group — Thiazide Treatment Group: Non-diabetics with sleep systolic blood pressure of 125-139 mm Hg and awake systolic blood pressure <160 mm Hg Participants will be treated with Indapamide 0.625mg once a day After 4 weeks of treatment, the investigators will monitor chemistries/electrolytes with a fingerstick point of care device and repeat ambulatory blood pressure monitoring the investigators will repeat ambulatory blood pressure monitoring at 4, 8, and 12 weeks after treatment initiation.
  If sleep systolic blood pressure is < 120 mm Hg, the investigators will continue treatment
  Arms: Thiazide Therapy Group
Drug: Intensified Thiazide Treatment Group — At 4 weeks of therapy, individuals initially assigned to the Thiazide treatment group whose ambulatory blood pressure recheck showed a sleep systolic blood pressure >120 mm Hg, the investigators will intensify their blood pressure medications by adding on Telmisartan 40 mg and Amlodipine 5 mg. In two week intervals, labs and ambulatory blood pressure will be measured. If the systolic blood pressure >120, then the doses of Telmisartan and Amlodipine will be up-titrated until the sleep systolic blood pressure is <120.
  Arms: Thiazide Therapy Group
Drug: Combination Medication Treatment Group — Combination Medication Treatment Group: Diabetics or sleep systolic blood pressure of ≥ 140 mm Hg, or awake systolic blood pressure of ≥ 160 mm Hg
  * Participants will be treated with starting doses of a long acting blood pressure regimen of Telmisartan 40 mg and Amlodipine 5 mg daily
  * After 2 weeks, the investigators will monitor chemistries/electrolytes with a fingerstick point of care device and repeat ambulatory blood pressure monitoring
    * If sleep systolic blood pressure is < 120 mm Hg, the investigators will continue treatment and repeat ambulatory blood pressure again in another 2 weeks to assess reproducibility
    * If sleep systolic blood pressure is > 120 mm Hg, the investigators will increase Telmisartan dose to 80 mg and the Amlodipine dose to 10 mg. Ambulatory blood pressure monitoring will be checked again after 2 weeks of therapy to verify efficacy.
  Arms: Combination Therapy Group

SUMMARY:
This is a protocol to obtain pilot data to submit a new NIH grant on Nocturnal Hypertension and Nocturia. In the diversity supplement to Dr. Victor's current NIH grant (Cut Your Pressure Too: The Los Angeles Barbershop Blood Pressure Study) the results show that uncontrolled systolic hypertension is an independent determinant of nocturia in African American men.

the investigators now want to pursue this correlation by designing a new NIH grant proposal to determine whether replacing short acting with long acting drugs and dosing them at bedtime rather than in the morning will: A. Lower systolic blood pressure during sleep B. Improve nocturia and result in better sleep quality

DETAILED DESCRIPTION:
Aims and Significance of pilot data

Determine:

1. The feasibility of the Southern California Healthy Heart and Blood Pressure registry as an effective method to recruit African American men to participate in a new research program
2. If participants are willing to comply with the study procedures including wearing an activity monitor, sleep study device, and ambulatory blood pressure monitor
3. The within subject variation for repeated measures of nocturnal blood pressure by ambulatory blood pressure and activity monitoring
4. If nocturnal systolic blood pressure is higher in men with self-reported nocturia ≥2 than in men with 0-1 nocturia
5. If use of long-acting antihypertensive medication as well as nighttime dosing of medication can lower nocturnal systolic blood pressure and reduce nocturia

Purpose:

Obtain key pilot data to show feasibility and document the reproducibility of the proposed measurements.

ELIGIBILITY:
Inclusion Criteria:

* African American Men
* Age 35 to 59 years-old
* Able to give informed consent
* Willing to wear the activity monitor, ambulatory blood pressure monitoring (ABPM), and sleep study device
* Uncontrolled hypertension: both a sleeping average systolic blood pressure of ≥ 125 mm Hg and an awake average systolic blood pressure of ≥ 135 mm Hg

Exclusion Criteria:

* Severe Sleep Apnea (Apnea Hypopnea Index (AHI) of > 30 on home sleep study) or history of sleep apnea diagnosis and use of Continuous Positive Airway Pressure therapy
* Uncontrolled Diabetes Mellitus (a random glucose of ≥ 200 mg/dL)
* History of diagnosis or symptoms of either prostate disease or overactive bladder (urinary urgency or frequency during the daytime)
* Chronic kidney disease (Glomerular filtration rate of < 60 mL/min/1.73 m2 based on the MDRD equation)
* Renal transplant recipient
* Loop diuretic use
* Night shift work
* On chemotherapy for cancer
* Orthostatic hypotension

  o After 2 minutes of standing: a drop in blood pressure of > 20/10 mm Hg, a standing systolic blood pressure of < 100 mm Hg, or tachycardia with an increased heart rate of > 20 beats/minute
* Other reasons deemed unsafe for study participation by Principle Investigator

Ages: 35 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Participant Compliance | 12 weeks
  If participants are willing to comply with the study procedures including wearing an activity monitor (it is built in the ambulatory blood pressure monitor), sleep study device, and ambulatory blood pressure monitor
change in the systolic blood pressure in participants | Change from Baseline Systolic Blood Pressure at 12 weeks
  The within subject variation in millimeter of mercury for repeated measures of nocturnal systolic blood pressure by ambulatory blood pressure.
change nocturnal systolic blood pressure in relation with frequency of nocturia | change from baseline at 12 weeks after treatment initiation.
  measurement of nocturnal systolic blood pressure will occur with continuous ambulatory blood pressure monitors. nocturia frequency will be self reported by participant and then verified by activity monitor (actigraph) built in the ambulatory blood pressure monitor .
Night time blood pressure medication dosing in relation with frequency of Nocturia | Change of systolic blood pressure from baseline at 12 weeks.
  the use of long-acting antihypertensive medication as well as nighttime dosing of medication can lower nocturnal systolic blood pressure and reduce the frequency of nocturia which will be self reported by participant and then verified by activity monitor (actigraph) built in the ambulatory blood pressure monitor .

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No